CLINICAL TRIAL: NCT06149910
Title: Evaluating the Uptake and Utility of Clinical Pathways for Newly Diagnosed Patients With Multiple Myeloma That Aim to Achieve and Maintain Measurable Residual Disease (MRD)-Negativity in Community Oncology Settings
Brief Title: Evaluating the Uptake and Utility of Clinical Pathways for Newly Diagnosed Patients With Multiple Myeloma
Status: Recruiting | Type: Observational
Sponsor: All4Cure (Industry)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: All4Cure03
Record Dates: First submitted 2023-11-17; First posted 2023-11-29 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma; Multiple Myeloma Without Mention of Remission
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Platform: Patients in this cohort are participating in the All4Cure platform and there has been an established intention to treat according to the clinical pathway. Additionally, the patient's primary physician will also be a participant in the All4Cure platform.
  Interventions: Other: Multiple Myeloma Pathway; Other: All4Cure Platform
- Documentation: Patients in this cohort are not participating in the All4Cure platform but there has been an established intention to treat according to the clinical pathway.
  Interventions: Other: Multiple Myeloma Pathway; Other: Documentation Pathway
- Off-pathway: Patients in this cohort are not participating in the All4Cure platform and there has not been in intention to treat according to the clinical pathway that has been established by a landmark time period.

INTERVENTIONS:
Other: Multiple Myeloma Pathway — Use and adherence to a multiple myeloma pathway.
  Groups: Documentation; Platform
Other: All4Cure Platform — Participant in the All4Cure platform.
  Groups: Platform
Other: Documentation Pathway — Use of multiple myeloma pathway through written documentation.
  Groups: Documentation

SUMMARY:
All4Cure is partnering with community oncology practices participating in the Quality Cancer Care Alliance (QCCA) and Exigent Research to develop a clinical pathway that standardizes the evaluation, treatment and ongoing management of patients with newly diagnosed multiple myeloma who wish to achieve and maintain MRD negativity.

This is a longitudinal retrospective study that will collect data from three separate cohorts of patients with newly diagnosed multiple myeloma (NDMM). The cohorts classify patients based on whether care is delivered under an intention to adhere to an MRD-targeted clinical pathway, and if so, whether the implementation of that clinical pathway occurs through participation in the All4Cure platform vs. through written documentation. The three cohorts are labeled: Platform, Documentation, and Off-Pathway.

DETAILED DESCRIPTION:
The study will employ two implementations of an MRD-targeted pathway one that disseminates pathway guidance through written documentation, and another that leverages the All4Cure platform to support pathway adherence through direct engagement of other experts, and through integration of elements of the MRD-targeted pathway into the structured components of the platform. The study also includes a comparator cohort of patients not being treated according to the clinical pathway. Analysis under the primary objective will evaluate outcomes between patients being treated following written pathway documentation and patients being treated off pathway. The primary endpoints are the proportion of patients with achievement of VGPR or better (≥VGPR), and the proportion of patients with a CR or better (≥CR), within 12 months. Secondary endpoints include MRD negativity, pathway adherence, time to next treatment (TTNT), progression-free survival (PFS), overall survival (OS), and obstacles to getting daratumumab treatment. Sustained MRD negativity is an exploratory endpoint.

Data will be collected retrospectively, through stratified random sampling by race within cohort, with patients accrued over a 12-month period. All patients will be followed over time after accrual, with minimum available follow-up of 12 months. Accordingly, the estimated period from first accrual to last follow-up will be approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma

  * Diagnosis must occur on or after the formal launch of the MRD-targeted clinical pathway in the Exigent network
  * Diagnosis must be indicated by the presence of any of the following diagnostic codes for multiple myeloma: [C90.00]
  * Diagnosis must be confirmed on human review of the medical record
* Age ≥ 18 years at qualifying diagnosis.
* Patient has continued to receive care at a QCCA/Exigent Research practice for at least 90 days after the index date.

Patients in the Documentation Cohort must meet the following additional inclusion criteria.

• Evidence in the record of a threshold level of adherence to the clinical pathway, or implied intention to adhere to the clinical pathway.

In addition to the inclusion criteria for the documentation cohort, patients in the Platform Cohort must meet the following additional inclusion criteria.

* A record of registration by the patient for participation in the All4Cure platform, including signed HIPAA release forms that allow All4Cure to access their medical records.
* A record of registration by the patient's primary treating physician for participation in the All4Cure platform.

Exclusion Criteria:

* Patients with a concurrent other malignancy (except basal cell carcinoma, squamous cell carcinoma of the skin, or in situ malignancies of breast or cervix), or those who have received treatment of another malignancy within three years prior to diagnosis of multiple myeloma (except for treatment of basal cell carcinoma, squamous cell carcinoma of the skin, or in situ malignancies of breast or cervix), are excluded from eligibility.
* Patients with multiple myeloma subtypes Immunoglobulin D (IgD) or Immunoglobulin E (IgE) are excluded due to the very low rate of these subtypes.
* Patients who transfer their care to another facility outside the QCCA/Exigent Research network within the first 90 days after NDMM diagnosis are excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients seen in a community oncology setting.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
To compare rate of tumor response and complete tumor response (≥VGPR and ≥CR) within 12 months of start of front-line therapy between the Documentation and Off-Pathway COHORT groups. | 24 months
  Tumor response will be a binary classification indicating the best tumor response documented through 12 months following start of front-line therapy, based on response assessment of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), stable disease (SD), progressive disease (PD) and not evaluable / not evaluated (NE). Given that the standard of care is to achieve at least a VGPR in the frontline setting, VGPR + sCR + CR will be defined as a tumor response, and other values will be interpreted as nonresponse for the purpose of this objective. Separately, sCR + CR will be interpreted as a complete tumor response, and other values will be interpreted as incomplete (VGPR) or nonresponse (PR, SD or PD). The proportion of patients who achieve VGPR or better any point within 12 months, and separately the proportion of patients who achieve a CR or better, will be compared between the Documentation and Off-Pathway COHORT groups.

SECONDARY OUTCOMES:
To compare pathway adherence between the Platform and Documentation COHORT group implementations of the MRD-targeted clinical pathway. | 24 months
  Pathway adherence will be quantified based on the adherence score, which reflects a sum of points credited for pathway-specified activities that are carried out during the 12-month period beginning from the start of treatment. The adherence score will be calculated at 3, 6 and 12-month periods with a minimum possible score of 0 points during all time periods. The maximum possible score will be 30 points during the 3 and 6-month time points and a maximum possible score of 40 points during the 12-month time point. The higher point scores indicate more adherence to the pathway.
To compare rate of tumor response and complete tumor response (≥VGPR and ≥CR) within 12 months of start of front-line therapy between PATHWAY groups (On-Pathway vs. Off-Pathway). | 12 months
To compare rate of tumor response and complete tumor response (≥VGPR and ≥CR) within 12 months of start of front-line therapy between the Platform and Off-Pathway COHORT groups. | 12 months
: To compare rate of tumor response and complete tumor response (≥VGPR and ≥CR) within 12 months of start of front-line therapy between the Documentation and Off-Pathway COHORT groups. | 12 months
  This will exclude Off-Pathway patients who received daratumumab as part of their front-line regimen.
To assess rates of MRD negativity (at 10-5 and 10-6 thresholds) at any point through 12 months after start of front-line therapy between the Platform and Documentation COHORT group implementations of the MRD-targeted clinical pathway. | 12 months
  MRD negativity will be assessed separately based on 10-5 (1/100,000) and 10-6 (1/1,000,000) thresholds, with rates of MRD negativity compared across the Platform and Documentation COHORT groups for each MRD negativity endpoint.
  Indication of MRD negativity at any point within 12 months of start of front-line therapy under each of the thresholds will be deemed to constitute MRD-negative status for that threshold endpoint, irrespective of evidence of MRD-positive status at other assessments.
To compare progression-free survival (PFS), time to next treatment (TTNT), and overall survival (OS) between the Documentation and Off-Pathway COHORT groups. | 12 months
  This will be done from a landmark at 6 months after start of front-line therapy, and to compare PFS, TTNT, and OS between the Platform and Documentation COHORT groups from that same landmark time point.
  To assess the sensitivity of the results to the selection of landmark timepoint, the analysis will also evaluate outcomes as measured from 3-month and 12-month landmarks.
To describe the frequency of patients that encountered obstacles reported in the record to accessing D-RVd for induction therapy or for accessing Dara-R for maintenance therapy from third-party payers. | 24 months
  If more than one obstacle type is reported per patient, each that is documented in the record will be endorsed.
  The frequency of patients who encountered each obstacle type, and the frequency of patients who encountered any obstacle (i.e., at least one obstacle), will be reported from among patients whom the record indicates attempted to get treatment with Daratumumab, Revlimid, Velcade, Dexamethasone (D-RVd) or Daratumumab, Revlimid (Dara-R), by COHORT group.
To describe the percentage of patients that encountered obstacles reported in the record to accessing D-RVd for induction therapy or for accessing Daratumumab, Revlimid (Dara-R) for maintenance therapy from third-party payers. | 24 months
  If more than one obstacle type is reported per patient, each that is documented in the record will be endorsed.
  The percentage of patients who encountered each obstacle type, and the percentage of patients who encountered any obstacle (i.e., at least one obstacle), will be reported from among patients whom the record indicates attempted to get treatment with Daratumumab, Revlimid, Velcade, Dexamethasone (D-RVd) or Daratumumab, Revlimid (Dara-R), by COHORT group.
To estimate the percentage of all patients with NDMM to whom care was provided within the QCCA/Exigent network from the date of the first patient enrolled to the date of the last patient enrolled. | 24 months
  This objective requires analysis of the enrolled patient sample as a subset of the underlying eligible population within the QCCA/Exigent network, and will be conducted through analysis of case screening data, without formal data collection from the underlying population of unaccrued eligible patients.

OTHER OUTCOMES:
To examine the rate of tumor response and complete tumor response (≥VGPR and ≥CR) within 12 months of the start of front-line therapy as a function of pathway adherence, controlling demographic and clinical characteristics. | 24 months
  * This exploratory objective considers the possibility that some patients and providers for whom there is a documented intent to adhere to the clinical pathway may not adhere very well, and this may attenuate the observed difference between the Documentation and Off-Pathway cohorts. If this occurs, analysis under this objective should isolate the effect of adherence more directly.
  * Note that analysis under this objective is not considered a substitute for cohort comparisons, because measurement of adherence in this study will be limited to a set of indicators that are likely to be documented in the electronic medical record (EMR).
To describe the rates of sustained MRD negativity (at 10-5 and 10-6 thresholds) observed during the study period across the Platform and Documentation COHORT group implementations of the MRD-targeted clinical pathway. | 24 months
  * Sustained MRD negativity will be defined as evidence of MRD negativity (at 10-5 and 10-6 thresholds) at least 6 months after a previous finding of MRD negativity, without an intervening finding of MRD positivity.
  * Note that patients will have variable durations of follow-up, and variable opportunity for observation of sustained MRD negativity. Consequently, this analysis under this objective will be descriptive only.
This exploratory objective will consider whether it is of interest to explore further analysis under those objectives with the subset of patients who are transplant eligible. | 24 months
  Specifications of the research questions for this subset would be as stated under each of the Objectives 1 through 7, above.

CONTACTS AND LOCATIONS:
Locations (1):
- All4Cure, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No